CLINICAL TRIAL: NCT04666272
Title: Effectiveness and Safety of Dabrafenib in Combination With Trametinib as Adjuvant Treatment for Chinese Patients With Stage III BRAF V600 Mutation-positive Melanoma After Complete Resection
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436FCN01
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: BRAF V600 mutation-positive melanoma; cutaneous or mucosal melanoma; China; dabrafenib; trametinib
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- dabrafenib in combination with trametinib as adjuvant treatment: Patients will be treated according to the China package insert for dabrafenib and trametinib. The approved starting doses of dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) will be used.
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — There is no treatment allocation. Patients administered dabrafenib alone by prescription that have started before inclusion of the patient into the study could be enrolled.
Drug: trametinib — There is no treatment allocation. Patients administered trametinib alone by prescription that have started before inclusion of the patient into the study could be enrolled.

SUMMARY:
This is a prospective, open label, single-arm, multicenter, non-interventional study of dabrafenib in combination with trametinib as adjuvant treatment for Chinese patients with stage III BRAF V600 mutation positive melanoma after complete resection.

DETAILED DESCRIPTION:
The study will consist of a treatment phase and follow-up phase. The treatment period is 12 months. Discontinuation of study treatment may occur earlier than 12 months for disease recurrence, death, unacceptable toxicity or withdrawal of consent. Patients will be followed for disease recurrence every 6 months and up to 24 months after the end of treatment (EOT)

ELIGIBILITY:
Inclusion Criteria:

Patient(s) must meet all of the following criteria to be eligible for inclusion:

1. ≥18 years old of age at the time of informed consent and of Chinese descent
2. Signed written informed consent
3. Going to receive commercial dabrafenib and trametinib according to approved label
4. Completely resected histologically confirmed Stage III BRAF V600 mutation positive cutaneous or mucosal melanoma as defined by the following staging systems:

   * for stage III cutaneous melanoma: as per American Joint Committee on Cancer (AJCC) 8th edition for melanoma
   * for stage III mucosal melanoma of the head and neck origin: as per AJCC 8th edition for mucosal melanoma of the head and neck
   * for stage III mucosal melanoma of anal canal, rectum and genital track origin: as per Chinese guidelines on the diagnosis and treatment of melanoma 2019 edition
5. Must be surgically rendered free of disease (defined as the date of the most recent surgery) no more than 12 weeks before enrollment
6. Recovered from definitive surgery (e.g. no uncontrolled wound infections or indwelling drains)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1

Exclusion Criteria:

Patient will be excluded from this study if he/she meets any of the following criteria:

1. Known ocular melanoma
2. Patient received other systemic neo-adjuvant and/or adjuvant therapy for melanoma (including dabrafenib in combination with trametinib started before ICF signature)
3. Patient is not able to comply with the planned study procedures
4. Taken an investigational drug within 28 days prior to enrolment
5. History of another malignancy (including melanoma) or a concurrent malignancy, except malignancies that were treated curatively and have not recurred within 2 years prior to treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include Chinese patients with stage III BRAF V600 mutation positive melanoma treated with dabrafenib in combination with trametinib in a commercial setting.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-12-31 (Actual); Primary Completion 2028-02-04 (Estimated); Study Completion 2028-02-04 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) | Up to 36 months
  Relapse-free survival (RFS), defined as the time from start of treatment to disease recurrence or death due to any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 36 months
  Overall survival (OS) defined as the time from start of treatment to death due to any cause
Safety of dabrafenib in combination with trametinib | Up to 36 months
  Adverse events (AEs) and serious adverse events (SAEs) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- China (9):
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing

IPD SHARING:
Plan to Share IPD: No